CLINICAL TRIAL: NCT00714246
Title: Phase I/II Study of Bortezomib (PS-341) in Combination With Carboplatin and Docetaxel for Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Bortezomib (PS-341) in Combination With Carboplatin and Docetaxel for Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Chandra P. Belani, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSU 26983
Record Dates: First submitted 2008-07-07; First posted 2008-07-14 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: advanced non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (7):
- Phase I - Dose Level 1 (Experimental): Carboplatin AUC 5 mg/ml/min (Day 1) Docetaxel 60 mg/m2 (Day 1) Bortezomib 0.7 mg/m2 (Day 1,4,8,11)
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Docetaxel
- Phase I - Dose Level 2A (Experimental): Carboplatin AUC 6 mg/ml/min (Day 1) Docetaxel 60 mg/m2 (Day 1) Bortezomib 0.7 mg/m2 (Day 1,4,8,11)
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Docetaxel
- Phase I - Dose Level 2B (Experimental): Carboplatin AUC 6 mg/ml/min (Day 1) Docetaxel 60 mg/m2 (Day 1) Bortezomib 1.0 mg/m2 (Day 1,4,8,11)
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Docetaxel
- Phase I - Dose Level 3 (Experimental): Carboplatin AUC 6 mg/ml/min (Day 1) Docetaxel 60 mg/m2 (Day 1) Bortezomib 1.0 mg/m2 (Day 1,4,8,11)
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Docetaxel
- Phase I - Dose Level 4 (Experimental): Carboplatin AUC 6 mg/ml/min (Day 1) Docetaxel 75 mg/m2 (Day 1) Bortezomib 1.0 mg/m2 (Day 1,4,8,11)
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Docetaxel
- Phase I - Dose Level 5 (Experimental): Carboplatin AUC 6 mg/ml/min (Day 1) Docetaxel 75 mg/m2 (Day 1) Bortezomib 1.3 mg/m2 (Day 1,4,8,11)
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Docetaxel
- Phase II (Experimental): Carboplatin AUC 5 mg/ml/min (Day 1) Docetaxel 60 mg/m2 (Day 1) Bortezomib 0.7 mg/m2 (Day 1,4,8,11)
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Bortezomib — Dose escalation using traditional Phase I - 3 x 3 design to establish MTD of bortezomib when administered in combination with carboplatin and docetaxel
  Other Names: VELCADE; PS-341
Drug: Carboplatin — Establish MTD of bortezomib when administered in combination with carboplatin and docetaxel
  Other Names: Paraplatin
Drug: Docetaxel — Establish MTD of bortezomib when administered in combination with carboplatin and docetaxel
  Other Names: Taxotere

SUMMARY:
This is a phase I/II study. The phase I portion of the study will determine the maximum tolerated dose of bortezomib when administered in combination with carboplatin & docetaxel and to determine the efficacy of the combination for patients with advanced NSCLC. Phase II will utilize the dosage determined in the Phase I and implement regimen to determine time to progression, overall survival, and changes in serum proteomics patterns before & after combination therapy.

DETAILED DESCRIPTION:
A chemotherapy efficacy plateau' has been reached for the treatment of patients with advanced or metastatic non-small cell lung cancer. Platinum-based two-drug combination is considered the current standard of care for the treatment of advanced NSCLC. There is a need to develop novel regimens to improve the outcome for patients with advanced NSCLC. The combination of carboplatin and docetaxel is effective for therapy of advanced NSCLC. This combination results in improved survival and quality of life for patients with advanced NSCLC. Docetaxel exhibits preclinical synergy with bortezomib.

The trial was intended to be a phase I/II study to define the maximum tolerated dose of bortezomib that can be administered in combination with docetaxel and carboplatin and subsequently evaluate the efficacy of the regimen for patients with advanced NSCLC. However, the trial never moved past the phase I portion of the study and was terminated early.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed stage IIIB (pleural or pericardial effusion) or stage IV NSCLC
* Age > 18 years
* ECOG PS < 2
* No prior chemotherapy
* Measurable disease
* Signed informed consent
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function

Exclusion Criteria:

* Untreated clinically active brain metastasis
* Radiotherapy within 2 weeks prior to initiation of protocol therapy
* Treatment with any investigational therapy within 4 weeks prior to enrollment
* History of any cancer other than NSCLC (except non-melanoma skin cancer or carcinoma on situ of the cervix) within the last 5 years
* Patients in their reproductive age group should use an effective method of birth control. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter. Patients who are breast-feeding will be excluded from the study. Women of childbearing potential must have a negative pregnancy test.
* Major surgery within 3 weeks prior to enrollment
* Use of immunosuppressive agents including systemic corticosteroids within 4 weeks prior to enrollment (corticosteroids are permitted as physiological replacement therapy or as supportive care for nausea and emesis)
* Known history of Human immunodeficiency virus infection
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the investigator
* Concurrent serious medical infection or illness, or psychiatric illness likely to interfere with participation in this clinical study.
* History of known hypersensitivity to docetaxel or other drugs formulated with polysorbate 80, bortezomib, boron or mannitol
* Patient has Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose of bortezomib when administered in combination with carboplatin & docetaxel for treatment of patients with advanced NSCLC cancer. Determine the response rate of the combination for patients with advanced NSCLC. | Expected average of 2 years

SECONDARY OUTCOMES:
Define dose-limiting toxicities of the combination of carboplatin, docetaxel & bortezomib for patients with advanced NSCLC. Determine the time to progression & overall survival, assess toxicities, determine changes in serum proteomics patterns | Expected average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P. Belani, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No